CLINICAL TRIAL: NCT02570919
Title: Phase II Randomized Study Comparing Ultra-high-dose Hypofractionated vs. Single-dose Image-Guided Radiotherapy (IGRT) With Urethral Sparing for Intermediate Risk Prostate Cancer
Brief Title: Phase II Study of Ultra-high-dose Hypofractionated vs. Single-dose Image-Guided Radiotherapy for Prostate Cancer
Acronym: PROSINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Carlo Greco, MD, M.D., Fundacao Champalimaud
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROSINT-IGRT A(1)
Record Dates: First submitted 2015-09-02; First posted 2015-10-07 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: PROSTATE CANCER
Keywords: Prostate cancer; IGRT; Hypofractionation; Extreme; Single Fraction; Urethral Sparing; MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IGRT 45 Gy in 5 fractions of 9 Gy (Active Comparator): Arm A: Hypofractionated IGRT at a prescription dose of 45 Gy in 5 fractions of 9 Gy delivered in five consecutive days
  Interventions: Radiation: IGRT 45 Gy in 5 fractions of 9 Gy
- IGRT 24 Gy single dose (Experimental): Arm B: single fraction IGRT at a prescription dose of 24 Gy
  Interventions: Radiation: IGRT 24 Gy single dose

INTERVENTIONS:
Radiation: IGRT 45 Gy in 5 fractions of 9 Gy — Administration of 9 Gy in five consecutive days, to a total dose of 45 Gy radiation
  Arms: IGRT 45 Gy in 5 fractions of 9 Gy
Radiation: IGRT 24 Gy single dose — Administration of a single dose of 24 Gy in one session
  Arms: IGRT 24 Gy single dose

SUMMARY:
The present study evaluates clinical outcomes and treatment-related toxicity following definitive ultra-high dose external beam radiotherapy delivered with two different regimens in patients with intermediate-risk adenocarcinoma of the prostate. Modern computer-driven technology enables the implementation of ultra-high hypofractionated Image-Guided Radiotherapy (IGRT) safely.

Prostate cancer patients classified according to the current National Comprehensive Cancer Network (NCCN) guidelines as intermediate risk (biopsy Gleason score of 7 and/or Prostate Specific Antigen (PSA) level >10 and ≤20 ng/mL and/or Stage T1, T2a, T2b or T2c) are eligible for this study.

Patients will undergo IGRT with volumetric intensity-modulated arc radiotherapy (VMAT) with state-of-the-art treatment-planning and quality assurance procedures. Emphasis is placed on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. A rectal balloon with air filling will be used for prostate target immobilization and anatomical reproducibility, while a urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking. Previously untreated patients with intermediate-risk prostate cancer will be prospectively randomized to receive either 45 Gy in five fractions of 9 Gy each vs. 24 Gy in a single-dose.

Patients will be followed at one month post-treatment and every 3 months for up to 12 months (+/- 4 weeks) and every 6 months thereafter. Acute and chronic toxicity evaluations will focus on urinary, rectal and sexual functions and will be assessed through validated questionnaires. Serum PSA values will be regularly acquired during follow-up. A multiparametric MRI will be performed at baseline, 6, 12 and 24 months following intervention. Additionally, a post-treatment diffusion-weighted MRI (DW-MRI) will be performed within 15 minutes of the first treatment, to measure early physiologic changes, such as perfusion and ischemia, that may correlate with clinically relevant end-points. Post-treatment prostate needle biopsies will be obtained at 24 months to evaluate pathologic response to therapy. The study will be continuously monitored for a minimum of 5 years. In the event unexpected severe (grade ≥3) toxicities are observed in any one of the treatment arms, the study will be terminated according to the stopping rule >3/first 15 patients.

DETAILED DESCRIPTION:
The present phase II randomized study evaluates the clinical outcomes and potential treatment-related toxicity following definitive ultra-high dose per fraction external beam radiation therapy delivered with two different regimens in patients with intermediate-risk adenocarcinoma of the prostate. An emerging body of data suggests that extreme hypofractionated radiation schedules, which employ ultra-high dose per fraction (≥7 Gy) in a small number of fractions (≤5), appear equal or superior to conventionally-fractionated (1.8- 2.0 Gy/fraction) and moderately hypo-fractionated schemes (2.5-3.5 Gy/fraction) in terms of both tumor control and toxicity profiles. Modern computer-driven technology enables the implementation of ultra-high hypofractionated Image-Guided Radiotherapy (IGRT) safely.

Prostate cancer patients classified according to the current National Comprehensive Cancer Network (NCCN) guidelines as intermediate risk (biopsy Gleason score of 7 and/or Prostate Specific Antigen (PSA) level >10 and ≤20 ng/mL and/or Stage T1, T2a, T2b or T2c) are eligible for this study.

Extensive experience on extreme hypo-fractionation in prostate has been accrued over the past two years using organ stabilization by means of an endorectal balloon and urethral sparing technique with on-line target motion tracking. The standard dose prescription with this technique has been 45 Gy over 5 consecutive days.

Outcome data on intermediate risk patients treated with single dose external beam radiotherapy are not yet available, although experience on single dose High Dose Radiotherapy (HDR) brachytherapy in prostate cancer indicates similar clinical outcomes and toxicity profiles to external beam hypofractionated schedules. Experience with ultra-high single dose radiotherapy for bone and soft tissue oligometastatic prostate cancer has been consistently shown to locally control >90% prostate cancer lesions, clearly indicating sensitivity of prostate cancer tissue to this mode of cancer radiotherapy. Stage IV oligometastatic prostate cancer patients failing androgen deprivation therapy were treated according to current standard of care with single dose 24 Gy to all foci of detectable disease, including the radiation-naive intraprostatic lesions, with excellent early results, using the same technique employed in the hypofractionated setting. Overall, toxicity profiles have been thus far extremely favorable indicating the intermediate range safety of this technique when applied to whole prostate radiotherapy. These data suggest single dose therapy when properly employed is both safe and effective in managing intra-prostatic cancer settings. Taken together, these observations provide the basis for the present prospective phase II study. Patients enrolled in the study will undergo image-guided, volumetric intensity-modulated arc radiotherapy (VMAT) with state-of-the-art treatment-planning and quality assurance procedures with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. A rectal balloon with air filling will be used for prostate target immobilization and anatomical reproducibility, while a urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking. Previously untreated patients with intermediate-risk prostate cancer will be prospectively randomized to receive either 45 Gy in five fractions of 9 Gy each vs. 24 Gy single-dose radiotherapy.

Patients will be followed at one month post-treatment and every 3 months for up to 12 months (+/- 4 weeks) and every 6 months thereafter. Acute and chronic toxicity evaluations will focus, though not exclusively, on urinary, rectal and sexual functions and will be assessed through validated questionnaires. Serum PSA values will be acquired with the same schedule as clinical follow-up. A multiparametric MRI will be performed at baseline, 6, 12 and 24 months following intervention. Additionally, a post-treatment diffusion-weighted MRI (DW-MRI) will be performed within 15 minutes of the first treatment. Post-treatment prostate core needle biopsies will be obtained once at 24 months to evaluate pathologic response to therapy.The purpose of this scan is to measure early physiologic changes, such as perfusion and ischemia, that may correlate with clinically relevant endpoints. The study will be continuously monitored for a minimum of 5 years. In the event unexpected severe (grade ≥3) toxicities are observed in any one of the treatment arms, the study will be terminated according to the standard stopping rule >3/first 15 patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed study specific informed consent form;
* Histologic confirmation of adenocarcinoma of the prostate by biopsy;
* PSA ≤ 20 ng/mL;
* Gleason score 7;
* Staging MRI must confirm American Joint Committee on Cancer (AJCC) stage T1, T2a, T2b or T2c;
* No direct evidence of regional or distant metastases after appropriate staging studies;
* Age ≥ 50;
* Performance Status 0-2;
* Internation Prostate Symptom Score score must be ≤ 15 (alpha blockers allowed);
* CT scan or Ultrasound-based volume estimation of prostate gland ≤ 100 grams;

Exclusion Criteria:

* Positive lymph-nodes or metastatic disease from prostate cancer on imaging studies
* Prior invasive malignancy unless disease-free for a minimum of 5 years
* Tumour Clinical stage T3 or T4 on MRI
* PSA > 20 ng/mL
* Gleason score > 7
* Previous pelvic radiotherapy
* Previous surgery for prostate cancer
* Previous transurethral resection of the prostate (TURP)
* History of Crohn's Disease or Ulcerative Colitis
* Previous significant urinary obstructive symptoms
* Significant psychiatric illness
* Ultrasound or CT estimate of prostate volume > 100 grams
* Severe, active co-morbidity

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by Common Toxicity Criteria for Adverse Effects v4.0 | Participants should be followed continuously, for the duration of 5 years
  Comparison of treatment related adverse events as measured by Common Toxicity Criteria for Adverse Effects v4.0 over a 5 year time frame

SECONDARY OUTCOMES:
Biochemical outcome based on PSA assessment | Participants should be followed at baseline and follow-up, for the duration of 5 years
Quality of life assessment based on validated questionnaires | Participants should be followed at baseline and follow-up, for the duration of 5 years
Pathological response based on biopsy at 24 months post-treatment | 24 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Greco, M.D., Principal Investigator — Champalimaud Foundation
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal

REFERENCES:
- [Derived] Greco C, Pares O, Pimentel N, Louro V, Santiago I, Vieira S, Stroom J, Mateus D, Soares A, Marques J, Freitas E, Coelho G, Seixas M, Lopez-Beltran A, Fuks Z. Safety and Efficacy of Virtual Prostatectomy With Single-Dose Radiotherapy in Patients With Intermediate-Risk Prostate Cancer: Results From the PROSINT Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 May 1;7(5):700-708. doi: 10.1001/jamaoncol.2021.0039. PMID 33704378
- [Derived] Bodo S, Campagne C, Thin TH, Higginson DS, Vargas HA, Hua G, Fuller JD, Ackerstaff E, Russell J, Zhang Z, Klingler S, Cho H, Kaag MG, Mazaheri Y, Rimner A, Manova-Todorova K, Epel B, Zatcky J, Cleary CR, Rao SS, Yamada Y, Zelefsky MJ, Halpern HJ, Koutcher JA, Cordon-Cardo C, Greco C, Haimovitz-Friedman A, Sala E, Powell SN, Kolesnick R, Fuks Z. Single-dose radiotherapy disables tumor cell homologous recombination via ischemia/reperfusion injury. J Clin Invest. 2019 Feb 1;129(2):786-801. doi: 10.1172/JCI97631. Epub 2019 Jan 14. PMID 30480549